CLINICAL TRIAL: NCT02323516
Title: Evaluation of the Efficacy of Low-dose Acetylsalicylic Acid on Diarrhea Induced by Anti-cancer Targeted Therapies.
Acronym: ASPIDIA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Ligue contre le cancer, France (Other); Canceropôle Nord Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ASPIDIA
Record Dates: First submitted 2014-11-19; First posted 2014-12-23 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Aspirin; Loperamide; Smectite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetylsalicylic acid + loperamide (Experimental): Acetylsalicylic acid + loperamide
  Interventions: Drug: diosmectite + loperamide
- diosmectite + loperamide (Active Comparator): Acetylsalicylic acid + loperamide
  Interventions: Drug: Acetylsalicylic acid + loperamide

INTERVENTIONS:
Drug: Acetylsalicylic acid + loperamide — In case of inefficiency in one month, according to predefined criteria, acetylsalicylic acid will be stopped and replaced by diosmectite.
  Arms: diosmectite + loperamide
Drug: diosmectite + loperamide — In case of inefficiency in one month, according to predefined criteria, diosmectite will be stopped and replaced by acetylsalicylic acid.
  Arms: Acetylsalicylic acid + loperamide

SUMMARY:
The mechanisms of action of the side effects associated with targeted therapies are still poorly understood. He was found in patients treated with gefitinib, increased levels of thromboxane B2 and P-selectin Thromboxane B2 is the result of the hydrolysis of thromboxane A2, which is itself obtained from Prostaglandin H2 under the action of the thromboxane synthetase. The thromboxane A2 is produced by platelets and the active pro-thrombotic properties as follows: stimulation of platelets and activation of other increased platelet aggregation.

The selectins are cell adhesion proteins with a role in the adhesion phenomena. P-selectin is expressed by platelets and endothelial cells.

The demonstration of increased plasma levels of thromboxane B2 and P-selectin leaves suggest a role of platelet activation in the occurrence of side effects associated with targeted therapies.

Kanazawa's study was conducted in 39 Japanese patients, trying to assess the value of low-dose acetylsalicylic acid or 100mg per day, that is to say, anti-aggrégantes doses, the occurrence rash and diarrhea induced by gefitinib.

In this study, the group of patients treated with acetylsalicylic acid presented a lower rate of side effects significantly, 58.3% versus 77.8%. The frequency of diarrhea was 18.5% (or 5 patients) in the standard group versus 0% in the group with acetylsalicylic acid. Similarly, it was found a reduction in the occurrence of skin rash, 33.3% or 4 patients in the acetylsalicylic acid group versus 74.1% s, 20 patients in the standard group. Finally, in this study, it was not revealed significant differences in terms of response to treatment with gefitinib (37% in the standard group versus 33% in the group treated with aspirin patient) It does not exist in our knowledge of prospective data evaluating the effect of acetylsalicylic acid on the reduction of side effects associated with targeted in a population of patients of Caucasian-type treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years old patient;
* WHO 0 to 2;
* Any solid tumor or hematologic malignancy requiring a tyrosine kinase inhibitor prescription in the absence of digestive disorders related to tumor disease;
* Treatment with one of the following targeted therapies: Gefitinib, erlotinib, sunitinib, sorafenib, Axitinib, Pazopanib, Lapatinib, Imatinib, afatinib,vemurafenib and Dabrafenib;
* Targeted therapy treatment whatever the processing line monotherapy, administered over a period of at least 15 days with continued dosing, with usual care recommendations;
* Diarrhea grade 1-3 according to NCI criteria CTCAE.4, in the absence of complications signs with at least 2 doses of loperamide per day.

Exclusion Criteria:

* Processing acetylsalicylic acid;
* Allergy or against-indications to acetylsalicylic acid (including concomitant antiplatelet or anticoagulant considered as increasing the risk of bleeding by the investigator) acid;
* Treatment with anti vitamin K or new oral anticoagulants;
* Absolute in pursuit of targeted therapy contraindication;
* Chronic diarrhea prior to clinical introduction of targeted therapy;
* Diarrhoea unrelated to targeted therapy such as:

  * extended resection of esophagus, inflammatory bowel disease, etc ...
  * carcinoid syndrome;
  * occlusive syndrome;
* Grade 3 diarrhea with signs of complications or grade 4
* Patients with a history of grade 3 diarrhea with signs of complications or grade 4 during previous treatment with TKI;
* Participation in other medical test;
* Pregnant women / nursing;
* Association with methotrexate at doses > 15 mg / d;
* Patient Trust or deprived of liberty.

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Efficacy measured by the decrease in the intensity of diarrhea and / or anti-diarrheal consumption | 1 month
  Effectiveness of acetylsalicylic acid versus diosmectite

SECONDARY OUTCOMES:
Toxicity | Three months
  Diarrhea decrease 3 months after the introduction of acetylsalicylic acid or diosmectite; Proportion of patients with a decrease in the grade of diarrhea during the months following the introduction of acetylsalicylic acid or diosmectite. Rate and intensity of side effects associated with other targeted therapy.
TKI dose reduction | Three months
  Proportion of patients requiring dose reduction of targeted therapy
Quality of life | Three months
  Quality of life and its evolution by month using ladders FACIT-G and FACIT-D.
Safety measured by the proportion of adverse event | Months 1 to 3
  Safety of acetylsalicylic acid in patients with diarrhea in targeted therapy

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHU, Amiens
  - Centre François Baclesse, Caen
  - Centre Hospitalier public du Cotentin, Cherbourg
  - Centre hospitalier, Compiègne
  - Centre Léon Bérard, Lyon